CLINICAL TRIAL: NCT04541004
Title: A 28-day, Single-armed, Open-label Trial to Evaluate Safety of the House Dust Mite (HDM) Sublingual Allergy Immunotherapy (SLIT) Tablet in Adolescent Subjects With HDM Allergic Rhinitis/Rhinoconjunctivitis With or Without Asthma
Brief Title: Adolescent Mite Allergy Safety Evaluation
Acronym: AMASE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ALK-Abelló A/S (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MT-18; 2020-000446-34 (EudraCT Number)
Record Dates: First submitted 2020-09-01; First posted 2020-09-09 (Actual); Results first posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2022-07

CONDITIONS: Allergic Rhinitis; Allergic Rhinoconjunctivitis
Keywords: Allergic rhinitis; House dust mite; Adolescent; Pediatric
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Intervention Model Description: single-armed
Masking Description: Non applicable
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HDM SLIT Tablet (Experimental): House dust mite (HDM) Sublingual allergy immunotherapy tablet
  Interventions: Biological: HDM SLIT-tablet

INTERVENTIONS:
Biological: HDM SLIT-tablet — Sublingual allergy immunotherapy tablet, for daily administration (1 tablet per day)
  Other Names: ACARIZAX, ODACTRA

SUMMARY:
This is a 28-day clinical trial studying the safety of the house dust mite tablet in adolescents with allergic rhinitis/rhinoconjunctivitis.

The purpose of this trial is to collect additional safety information about a tablet used to treat house dust mite allergies, when used to treat adolescents who have these allergies.

The trial medication used is already approved to treat allergic rhinitis caused by house dust mite in adults and adolescents (12-17 years old) in several countries.

DETAILED DESCRIPTION:
This trial is a 28-day, single-arm open-label phase III trial to evaluate safety of the house dust mite SLIT-tablet in adolescents (12-17 years of age) with HDM allergic rhinitis/rhinoconjunctivitis with or without asthma. Approximately 250 adolescents will be enrolled in the trial and will receive the house dust mite SLIT tablet. The trial is conducted in several European countries.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Male or female subjects aged ≥12 to ≤17 years
* A clinical history of allergic rhinitis/rhinoconjunctivitis (AR/C) when exposed to HDM
* Positive skin prick test (SPT) to Dermatophagoides pteronyssinus and/or Dermatophagoides farinae at screening
* Lung function measured by Forced expiratory volume in 1 second (FEV1) ≥ 70% of predicted value or according to local requirements while on subject's usual asthma medication
* The subject must be willing and able to comply with trial protocol and adhere to IMP treatment

Main Exclusion Criteria:

* A subject who has previously been included in studies with the HDM SLIT-tablet, or otherwise being treated with the marketed HDM SLIT-tablet (e.g. ACARIZAX, ODACTRA)
* Any SLIT or SCIT treatment with D. pteronyssinus or D. farinae reaching the maintenance dose within the last 5 years. In addition, any SLIT or SCIT treatment with D. pteronyssinus or D. farinae within the previous 12 months prior to visit 1
* Ongoing treatment with any allergy immunotherapy product at screening
* Severe chronic oral inflammation
* A diagnosis or history of eosinophilic oesophagitis
* Any clinical deterioration of asthma that resulted in emergency treatment, hospitalisation or treatment with systemic corticosteroids within 3 months prior to first tablet administration
* Female with positive urine pregnancy test, breastfeeding, pregnant or planning to become pregnant within the projected duration of the trial
* Sexually active female of childbearing potential without medically accepted contraceptive method

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 253 (Actual)
Dates: Start 2020-09-23 (Actual); Primary Completion 2021-04-24 (Actual); Study Completion 2021-04-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Horn, MD, Principal Investigator — HNO Praxis am Neckar
Locations (27):
- Czechia (8):
  - Alergologicka ambulance, Čáslav
  - Alergopraktik s.r.o., Jablonec nad Nisou
  - Allergology Jihlava, Jihlava
  - Oblastni nemocnice Kolin, a.s. Detske oddeleni. Alergologicka a, Kolín
  - Alergologicka ordinace, Kutná Hora
  - Alergomyšl s.r.o., Litomyšl
  - Alergologie SKOPKOVA s.r.o., Ostrava
  - KASMED s.r.o., Tábor
- Germany (7):
  - HNO Praxis am Neckar, Heidelberg, Baden-Wrttemberg
  - Praxis Dres. med. Florian Heimlich und Angelika Witzel-Heimlich, Heidelberg, Baden-Wurttemberg
  - Praxis Dr. Decot, Dreieich, Hesse
  - Kinderarztpraxis BramscheDr. Thomas Adelt, Bramsche, Lower Saxony
  - HNO-Praxis Dr. med. Udo Schaefer, Dresden, Saxony
  - Facharzt fr HNO und Allergologie, Dresden, Saxony
  - HNO-Genossenschaft Sachsen-Anhalt E.G., Wolmirstedt, Saxony-Anhalt
- Slovakia (12):
  - Ambulancia klinickej imunologie a alergologie, Banská Bystrica
  - ALIAN s.r.o., Bardejov
  - Jocia s.r.o., Bratislava
  - AlergoImuno centrum s.r.o. - Ambulancia alergologi, Kežmarok
  - ALERGO H2B s.r.o. Ambulancia klinickej imunológie a alergológie, Komárno
  - Alersa, Košice
  - Ambulancie klinickej imunologie a alergologie Univerzitna nemocnica Martin, Martin
  - NZZ Imunologicka ambulancia, Poprad
  - Alergo immunological center prešov, Prešov
  - Diagnosticke centrum - Ambulancia klinickej imunologie a alergologie, Zoll-Med, s.r.o., Rimavská Sobota
  - Ambulancia klinickej imunologie a alergologie, NZZ Ambulancia klinickej imunologie, Šurany
  - Medimun s.r.o., Trnava

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | HDM SLIT Tablet
Started | 253
Completed | 251
Not Completed | 2
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Arm/Group | HDM SLIT Tablet
Number analyzed (Participants) | 253
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 253
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101
  Male | 152
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 229
  Unknown or Not Reported | 18
Region of Enrollment [Count of Participants; unit: Participants]
  Czechia | 87
  Slovakia | 137
  Germany | 29
Height [Mean (Standard Deviation); unit: cm] | 166.3 (10.6)
Weight [Mean (Standard Deviation); unit: kg] | 61 (15.1)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 21.9 (4.38)
Smoking history [Count of Participants; unit: Participants]
  Current | 3
  Never | 250
Regularly exposed to tobacco smoke [Count of Participants; unit: Participants]
  No | 246
  Yes | 4
  Not applicable (current smokers) | 3
Baseline sensitisations [Count of Participants; unit: Participants]
  HDM only | 112
  HDM and others | 141
Duration of HDM allergic rhinitis/rhinoconjunctivitis [Mean (Standard Deviation); unit: years] | 5.9 (3.5)
Asthma status [Count of Participants; unit: Participants]
  No | 144
  Yes | 109
Inhaled corticosteroids [Count of Participants; unit: Participants]
  No | 180
  Yes | 73
Duration of asthma [Mean (Standard Deviation); unit: years] | 6.7 (3.9)
FEV1 (percentage predicted) [Mean (Standard Deviation); unit: percentage predicted FEV1] | 96.10 (12.84)
FEV1 (L) [Mean (Standard Deviation); unit: liters] | 3.26 (0.78)

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With at Least One Treatment-emergent Adverse Event (TEAE)
Description: At least one TEAE
Time Frame: From time of first IMP administration and no later than 7 days after last IMP administration, approximately 35 days.
Measure: Number; unit: subjects
Arm/Group | HDM SLIT Tablet
Number analyzed (Participants) | 253
subjects | 223

2. Primary Outcome: Proportion of Subjects With at Least One Treatment-emergent Adverse Event (TEAE)
Description: At least one TEAE
Time Frame: From time of first IMP administration and no later than 7 days after last IMP administration, approximately 35 days.
Measure: Number (90% Confidence Interval); unit: percent
Groups:
- HDM SLIT Tablet: House dust mite (HDM) Sublingual allergy immunotherapy tablet HDM SLIT-tablet: Sublingual allergy immunotherapy tablet, for daily administration (1 tablet per day)
Arm/Group | HDM SLIT Tablet
Number analyzed (Participants) | 253
percent | 88.1 [84.3 to 91.3]

3. Primary Outcome: Number of Treatment-emergent Adverse Events (TEAEs)
Description: At least one TEAE
Time Frame: From time of first IMP administration and no later than 7 days after last IMP administration, approximately 35 days.
Measure: Number; unit: events
Arm/Group | HDM SLIT Tablet
Number analyzed (Participants) | 253
events | 1940

4. Secondary Outcome: Number of Subjects With at Least One Solicited Treatment-emergent Adverse Event (TEAE)
Description: At least one solicited TEAE
Time Frame: From time of first IMP administration and no later than 7 days after last IMP administration, approximately 35 days.
Measure: Number; unit: subjects
Arm/Group | HDM SLIT Tablet
Number analyzed (Participants) | 253
subjects | 216

5. Secondary Outcome: Proportion of Subjects With at Least One Solicited Treatment-emergent Adverse Event (TEAE)
Description: At least one solicited TEAE
Time Frame: From time of first IMP administration and no later than 7 days after last IMP administration, approximately 35 days.
Measure: Number (90% Confidence Interval); unit: percent
Arm/Group | HDM SLIT Tablet
Number analyzed (Participants) | 253
percent | 85.4 [81.2 to 88.9]

6. Secondary Outcome: Number of Solicited Treatment-emergent Adverse Events (TEAEs)
Description: At least one solicited TEAE
Time Frame: From time of first IMP administration and no later than 7 days after last IMP administration, approximately 35 days.
Measure: Number; unit: events
Arm/Group | HDM SLIT Tablet
Number analyzed (Participants) | 253
events | 1796

7. Secondary Outcome: Number of Subjects With at Least One IMP-related Adverse Event (AE)
Description: At least one IMP-related AE
Time Frame: From time of first IMP administration and no later than 7 days after last IMP administration, approximately 35 days.
Measure: Number; unit: subjects
Arm/Group | HDM SLIT Tablet
Number analyzed (Participants) | 253
subjects | 218

8. Secondary Outcome: Proportion of Subjects With at Least One IMP-related Adverse Event (AE)
Description: At least one IMP-related AE
Time Frame: From time of first IMP administration and no later than 7 days after last IMP administration, approximately 35 days.
Measure: Number (80% Confidence Interval); unit: percent
Arm/Group | HDM SLIT Tablet
Number analyzed (Participants) | 253
percent | 86.2 [82.1 to 89.6]

9. Secondary Outcome: Number of IMP-related Adverse Events (AEs)
Description: At least one IMP-related AE
Time Frame: From time of first IMP administration and no later than 7 days after last IMP administration, approximately 35 days.
Measure: Number; unit: events
Arm/Group | HDM SLIT Tablet
Number analyzed (Participants) | 253
events | 1863

10. Secondary Outcome: Number of Subjects With At Least One Treatment-emergent Serious Adverse Event (SAE)
Description: At least one treatment-emergent SAE
Time Frame: From time of first IMP administration and no later than 7 days after last IMP administration, approximately 35 days.
Measure: Number; unit: subjects
Arm/Group | HDM SLIT Tablet
Number analyzed (Participants) | 253
subjects | 0

11. Secondary Outcome: Proportion of Subjects With At Least One Treatment-emergent Serious Adverse Event (SAE)
Description: At least one treatment-emergent SAE
Time Frame: From time of first IMP administration and no later than 7 days after last IMP administration, approximately 35 days.
Measure: Number (90% Confidence Interval); unit: percent
Arm/Group | HDM SLIT Tablet
Number analyzed (Participants) | 253
percent | 0 [0 to 1.18]

12. Secondary Outcome: Number of Treatment-emergent Serious Adverse Events (SAEs)
Description: At least one treatment-emergent SAE
Time Frame: From time of first IMP administration and no later than 7 days after last IMP administration, approximately 35 days.
Measure: Number; unit: events
Arm/Group | HDM SLIT Tablet
Number analyzed (Participants) | 253
events | 0

ADVERSE EVENTS:
Time Frame: AEs were collected from consent to 7 days after end-of-trial or discontinuation (from first IMP intake to 7 days after end-of-trial or discontinuation, up to 35 days).
Description: An AE is any untoward medical occurrence in a clinical trial subject, and which does not necessarily have a causal relationship with the administered IMP.
  An AE can therefore be any unfavourable and unintended sign (including e.g. a medication error), symptom, or disease, whether considered related to the IMP.
Arm/Group | HDM SLIT Tablet
All-Cause Mortality (participants affected / at risk) | 0/253
Serious Adverse Events (participants affected / at risk) | 0/253
Other Adverse Events (participants affected / at risk) | 223/253
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HDM SLIT Tablet (N=253)
Pharyngeal paraesthesia (Respiratory, thoracic and mediastinal disorders) | 17 (34)
Pharyngeal swelling (Respiratory, thoracic and mediastinal disorders) | 33 (59)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 132 (323)
Dysgeusia (Nervous system disorders) | 16 (24)
Ear pruritus (Ear and labyrinth disorders) | 101 (270)
Abdominal pain upper (Gastrointestinal disorders) | 40 (77)
Diarrhoea (Gastrointestinal disorders) | 24 (30)
Enlarged uvula (Gastrointestinal disorders) | 14 (38)
Glossodynia (Gastrointestinal disorders) | 41 (87)
Lip oedema (Gastrointestinal disorders) | 11 (15)
Lip swelling (Gastrointestinal disorders) | 40 (89)
Mouth swelling (Gastrointestinal disorders) | 14 (32)
Mouth ulceration (Gastrointestinal disorders) | 38 (68)
Nausea (Gastrointestinal disorders) | 40 (83)
Oedema mouth (Gastrointestinal disorders) | 21 (35)
Oral pain (Gastrointestinal disorders) | 10 (19)
Oral pruritus (Gastrointestinal disorders) | 169 (421)
Swollen tongue (Gastrointestinal disorders) | 29 (51)
Tongue eruption (Gastrointestinal disorders) | 6 (16)
Tongue ulceration (Gastrointestinal disorders) | 42 (79)
Vomiting (Gastrointestinal disorders) | 6 (9)
Rhinitis (Infections and infestations) | 6 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-08): https://cdn.clinicaltrials.gov/large-docs/04/NCT04541004/Prot_SAP_000.pdf